CLINICAL TRIAL: NCT04226898
Title: A Double-Blind Placebo-Controlled Trial of the Synbiotic Compound Probio-Tec ABCG for Schizophrenia Patients With and Without Elevated Markers of Gastrointestinal Inflammation
Brief Title: Synbiotic Compound to Reduce Symptoms of Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheppard Pratt Health System (Other)
Responsible Party: Principal Investigator, Faith Dickerson, Principal Investigator, Stanley Research Program, Sheppard Pratt Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMRI/SPHS: 2020-01
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Synbiotics; Synbiotic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Synbiotic Supplement (Experimental): The active synbiotic supplement consists of a stick/packet containing 4 strains of probiotic microorganisms: Lactobacillus acidophilus, LA-5® (material number 501082 FD LAK KGPharma); Lactobacillis paracasei subsp. paracasei, L. CASEI 431® (material number 684301 FD L. casei 431 HA Granulate); Lactobacillus rhamnosus, LGG® (material number 699817 FD LGG HA-W-IF); and Bifidobacterium animalis subsp. lactis, BB-12® (material number 699813 FD BB-12 HA-W-IF). In addition, the stick/sachet contains 5 g inulin. The product is a powder which participants will be asked to take with liquid or food. In this arm, the participant will take 1 powder stick of the synbiotic supplement once a day for 12 weeks after a 2-week placebo run-in.
  Interventions: Biological: Synbiotic Supplement
- Inert Compound (Placebo Comparator): The inert compound placebo looks identical to the synbiotic supplement. In this arm, the participant will take 1 powder stick of the placebo daily for 12 weeks after a 2 week placebo run-in.
  Interventions: Biological: Inert Compound

INTERVENTIONS:
Biological: Synbiotic Supplement — Synbiotic supplement 1 powder stick by mouth daily
  Other Names: Probio-Tec® ABCG-Stick-25
  Arms: Synbiotic Supplement
Biological: Inert Compound — Synbiotic supplement identical placebo 1 powder stick by mouth daily
  Arms: Inert Compound

SUMMARY:
The purpose of this study is to determine if taking a synbiotic supplement versus a placebo will reduce symptoms of schizophrenia when used in addition to standard antipsychotic medications.

DETAILED DESCRIPTION:
A total of n=68 participants with schizophrenia or schizoaffective disorder who have residual psychotic symptoms which are of at least moderate severity will be randomized. Intestinal inflammation will be assessed through the measurement of antibodies to Saccharomyces cerevisiae, gliadin, Candida albicans as well as high-sensitivity C-Reactive protein and Pentraxin-3. The duration of the trial is 14 weeks: after a 2-week placebo run in, the participants will be randomized to receive the synbiotic compound or identical-appearing placebo over the 12 weeks of the randomized phase. The synbiotic compound is a quality-tested product, Probio-Tec ABCG-Stick-25, manufactured by ChrHansen which contains 4 strains of probiotic microorganisms - Bifidobacteria BB-12, Lactobacillus casei, Lactobacillus acidophilus, and Lactobacillus rhamnosus - and the prebiotic, inulin, a fructan-containing polysaccharide which has been shown to increase the level of non-pathogenic bacteria in the gastrointestinal tract. All participants will also be maintained on a stable regimen of psychiatric medications prescribed by their treating psychiatrist.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, inclusive.
* Capacity for written informed consent.
* Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnosis of schizophrenia or schizoaffective disorder (APA 2013) as determined by the Structured Clinical Interview for DSM-5 Disorders (SCID-5).
* Outpatient at the time of enrollment.
* Residual psychotic symptoms of at least moderate severity as evidenced by a Positive and Negative Syndrome Scale (Kay et al., 1987) (PANSS) total score of 60 or higher AND one or more of the following: one or more PANSS positive symptom scores of 4 or higher; OR containing at least three positive or negative items with scores of 3 or higher at the screening visit.
* Receiving antipsychotic medication for at least 8 weeks prior to starting the study with no medication changes within the previous 21 days.
* Proficient in the English language.

Exclusion Criteria:

* DSM-5 diagnosis of intellectual disability or comparable diagnosis determined by previous versions of the DSM.
* Any clinically significant or unstable medical disorder as determined by the investigators, including congestive heart failure, liver disease, renal failure, any diagnosis of cancer undergoing active treatment.
* A primary immunodeficiency condition such as HIV infection, or undergoing cancer chemotherapy, or receiving systemic corticosteroids, methotrexate or monoclonal antibodies for treatment of an autoimmune disorder.
* History of IV drug use.
* DSM-5 diagnosis of a moderate or severe substance use disorder, except for caffeine or tobacco, within the last three months prior to the screening visit. If the patient has a positive drug toxicity screen at the time of visit 1 (screening) further evaluation by the investigator will be done of the substance use to determine eligibility.
* Participated in any investigational drug trial in the past 30 days.
* Pregnant or planning to become pregnant during the study period.
* Receipt of antibiotic medication within the 14 days prior to visit 2 (as anaerobic organisms residing in the gastrointestinal tract may be minimally affected by antibiotics). Of note, patients on antibiotic may be re-screened once the minimum duration of time since antibiotics use has been met.
* Current and regular use of a probiotic and or prebiotic supplement within the past 2 weeks. Of note, patients taking prebiotic or probiotic supplements may be re-screened.
* Documented inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis) or celiac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) Score From the Start to the End of the Double-blind Treatment Phase | 12 weeks (week 2 to week 14)
  The Positive and Negative Syndrome Scale (PANSS) measures psychiatric symptomatology, especially related to psychosis. The complete PANSS contains ratings for 30 symptoms, including 7 positive symptoms, 7 negative symptoms, and 16 general psychiatric symptoms. The severity of each symptom is rated on a scale ranging from 1 (minimal) to 7 (extreme); higher scores indicate increased symptomatology. Total PANSS scores include scores from all categories and range from 30 to 210 units on a scale.

SECONDARY OUTCOMES:
Change in the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) score from the start of the placebo run-in to the end of the double-blind phase | 14 weeks (week 0 to week 14)
  Cognitive performance is measured by the MATRICS Consensus Cognitive Battery composite score in participants. MCCB is comprised of 10 tests: Trail Making Test Part A; Brief Assessment in Cognition in Schizophrenia Symbol Coding; Hopkins Verbal Learning Test-Revised; Wechsler Memory Scale-III Spatial Span; Letter Number Sequencing; Neuropsychological Assessment Battery Mazes; Brief Visuospatial Memory Test-Revised; Category Fluency Animal Naming; Mayer-Salovey-Caruso Emotional Intelligence Test Managing Emotions; and Continuous Performance Test-Identical Pairs. For each test, a score is derived based on the raw item values. Each of the individual item raw scores is standardized to age and gender corrected tscores which are then summed to convert into a composite score ranging from <214->486 based on the MCCB scoring manual, with a higher score reflecting better performance.
Intestinal Inflammation Markers (#1) Antibodies to Saccharomyces cerevisiae | Screening, Week 8, Week 14
  Levels of intestinal inflammation will be assessed by the measurement of antibodies by immunoassays to Saccharomyces cerevisiae. (All of the immunoassays will be analyzed on the same scale. This is accomplished by standardizing the optical density values obtained from the immunoassays to those of a control population without a psychiatric disorder normalized to have a mean value of 1 and a standard deviation of 1. To adjust for multiple comparisons in the analysis of the 5 markers, the false discovery correction of Benjamani-Hochberg will be used.)
Intestinal Inflammation Markers (#2) Antibodies to Gliadin | Screening, Week 8, Week 14
  Levels of intestinal inflammation will be assessed by the measurement of antibodies by immunoassays to gliadin. (All of the immuoassays will be analyzed on the same scale. This is accomplished by standardizing the optical density values obtained from the immunoassays to those of a control population without a psychiatric disorder normalized to have a mean value of 1 and a standard deviation of 1. To adjust for multiple comparisons in the analysis of the 5 markers, the false discovery correction of Benjamani-Hochberg will be used.)
Intestinal Inflammation Markers (#3) Antibodies to Candida albicans | Screening, Week 8, Week 14
  Levels of intestinal inflammation will be assessed by the measurement of antibodies by immunoassays to Candida albicans. (All of the immunoassays will be analyzed on the same scale. This is accomplished by standardizing the optical density values obtained from the immunoassays to those of a control population without a psychiatric disorder normalized to have a mean value of 1 and a standard deviation of 1. To adjust for multiple comparisons in the analysis of the 5 markers, the false discovery correction of Benjamani-Hochberg will be used.)
Intestinal Inflammation Markers (#4) C-reactive protein | Screening, Week 8, Week 14
  Levels of intestinal inflammation will be assessed by the measurement of high-sensitivity C-reactive protein. (All of the immunoassays will be analyzed on the same scale. This is accomplished by standardizing the optical density values obtained from the immunoassays to those of a control population without a psychiatric disorder normalized to have a mean value of 1 and a standard deviation of 1. To adjust for multiple comparisons in the analysis of the 5 markers, the false discovery correction of Benjamani-Hochberg will b used.)
Intestinal Inflammation Markers (#5) Pentraxin-3 | Screening, Week 8, Week 14
  Levels of intestinal inflammation will be assessed by the measurement of Pentraxin-3. (All of the immunoassays will be analyzed on the same scale. This is accomplished by standardizing the optical density values obtained from the immunoassays to those of a control population without a psychiatric disorder normalized to have a mean value of 1 and a standard deviation of 1. To adjust for multiple comparisons in the analysis of the 5 markers, the false discovery correction of Benjamani-Hochberg will be used.)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Dickerson, PhD, MPH, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppard Pratt Health System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, symptom, and cognitive data will be shared with the National Database for Clinical Trials Related to Mental Illness (NDCT). Access may be obtained through an approved application with the NDCT.